CLINICAL TRIAL: NCT02142205
Title: A Prospective, Open-label, Non-randomized, Clinical Trial to Evaluate the Safety and Efficacy in RUSsian RRMS Patients on One Year Treatment With Natalizumab (TYSabri®).
Brief Title: Safety and Efficacy of Natalizumab (BG00002, Tysabri®) in Russian Participants With Relapsing Remitting Multiple Sclerosis (RRMS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RUS-TYS-11-10158
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BG00002 (natalizumab) (Experimental): 300 mg IV infusion every 4 weeks
  Interventions: Biological: BG00002

INTERVENTIONS:
Biological: BG00002 — IV Infusion
  Other Names: Tysabri®

SUMMARY:
The primary objective is to evaluate the safety and tolerability of natalizumab (BG00002, Tysabri®) in the study population (Russian participants with relapsing remitting multiple sclerosis). The secondary objectives are to look at evaluation of severity of relapse, hospitalization and steroid use requirement; Expanded Disability Status Scale (EDSS), functional tests, quality of life self-assessment questionnaires including the short form health survey self-assessment questionnaire (SF-36) and multiple sclerosis impact scale 29 (MSIS-29), evidence of MRI disease activity, participants free of disease activity (clinical activity and/MRI activity) and anti JC Virus (JCV) antibody evaluation.

ELIGIBILITY:
Key Inclusion Criteria:

* Must be natalizumab naïve.
* Must have a documented diagnosis of a relapsing remitting form of MS as defined by the revised McDonald Committee criteria (Polman et al., 2011)
* Must have had at least 1 relapse in the previous year:
* Must be stable in disability for at least 30 days prior to enrollment to the study
* Must be stable in symptomatic management of the disease, specifically spasticity, depression and fatigue for at least 30 days prior to enrollment to the study.
* Must be considered by the Investigator to be free of signs and symptoms suggestive of Progressive multifocal leukoencephalopathy (PML) based on medical history, physical examination, or laboratory testing.
* Must be willing to discontinue and remain free from concomitant immunosuppressive or immunomodulatory treatment (including IFN-beta and Glatiramer Acetate) while being treated with natalizumab during the study.

Key Exclusion Criteria:

Medical History:

* Onset of a relapse within 50 days prior to first infusion.
* Considered by the Investigator to be immunocompromised, based on medical history, physical examination, or laboratory testing or due to prior immunosuppressive treatment
* History of, or available abnormal laboratory results indicative of, any significiant viral, cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, gastrointestinal, dermatologic, psychiatric (including major depression), renal, and/or other major disease that would preclude the administration of a recombinant humanized antibody immunomodulating agent. The Investigator must re-review the subject's medical fitness for participation and consider any diseases that would preclude treatment.
* History of malignancy (subjects with basal cell carcinoma that has been completely excised prior to study entry remain eligible)
* Known history of human immunodeficiency virus infection or hematological malignancy
* History of organ transplantation (including anti-rejection therapy)
* A clinically significant infectious illness (e.g. abscess, pneumonia, septicemia) within 30 days prior to the Screening Visit.

Treatment History:

- Treatment with any kind of immunosuppressant medications (e.g., mitoxantrone, cyclophosphamide, cyclosporine, azathioprine, methotrexate, fingolimod, cladribine) within 6 months prior to Screening

Miscellaneous:

* Female subjects who are not postmenopausal for at least 1 year, surgically sterile (does not include tubal ligation), or unwilling to practice effective contraception (as defined by the Investigator) during the study
* Women who are breastfeeding, pregnant, or planning to become pregnant while on study
* Other unspecified reasons that, in the opinion of the Investigator and/or Biogen Idec, make the subject unsuitable for enrollment into this study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of participants that experience Serious Adverse Events (SAEs) and adverse events (AEs) | Up to Week 52

SECONDARY OUTCOMES:
Annualized relapse rate (ARR) | Up to Week 52
Time course to first relapse | Up to Week 52
Severity of relapse as measured by the Number of relapses requiring hospitalization and the Number of relapses requiring steroid treatment | Up to Week 52
Number of participants that do not experience a relapse | Up to Week 52
Change in EDSS scores | Up to Week 48
Duration of time to progression as measured by EDSS score | Up to Week 48
Number of participants that do not experience a progression in EDSS score | Up to Week 48
Percentage of participants with improvement in EDSS scores | Up to Week 48
  Measured by at least 1.0 point for 3 months sustained for participants with EDSS greater than or equal to, 2 at baseline
Changes from baseline in nine hole peg test (9HPT) | Up to Week 48
  A brief, standardized, quantitative test of upper extremity function. Both the dominant and non-dominant hands are tested twice. The participant is seated at a table with a small, shallow container holding 9 pegs and a wood or plastic block containing 9 empty holes. On a start command when a stopwatch is started, the partipant picks up the 9 pegs one at a time as quickly as possible, puts them in the 9 holes, and, once they are in the holes, removes them again as quickly as possible one at a time, replacing them into the shallow container. The total time to complete the task is recorded
Changes in Timed 25 foot walk from baseline | Up to Week 48
  A quantitative mobility and leg function performance test based on a timed 25-walk. It is the first component of the Multiple Sclerosis Functional Composite (MSFC) to be administered at each visit. The participant is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the participant has reached the 25-foot mark. The task is immediately administered again by having the participant walk back the same distance. Assistive devices may be used
Changes in cognition as assessed by the Symbol digit modalities test (SDMT) | Up to Week 48
  A simple substitution task that gives the examinee 90 seconds to pair specific numbers with given geometric figures. Examinees can give either written or spoken responses, making the test well suited for use with individuals who have motor disabilities or speech disorders. Because it involves only geometric figures and numbers, the SDMT is relatively free of cultural bias and can be administered to individuals who do not speak English.
Changes from baseline in visual function test (VFT) | Up to Week 48
Impact on participants quality of life using SF-36 and MSIS-29 self-assessment questionnaires | Up to Week 48
Percentage of participants that do not experience a relapse or progression in EDSS score | Month 12
Number of T1 gadolinium (Gd) enhancing lesions | At Week 48
Number of new T2 hyper intense lesions | At Week 48
  Compared to baseline
Number of newly enlarging T2 hyper intense lesions | At Week 48
  Compared to baseline
Number of new hypo intense T1 lesions (black holes) | At Week 48
Number of conversion of Gd lesions into black holes | At Month 12
Percentage of participants that do not experience a relapse as measured by an EDSS score that is not indicative of progression | At Month 12
Percentage of participants that do not develop new GD+ and new or newly enlarging T2 hyper intense lesions | At Week 48
Proportion of participants free of disease activity: no clinical & no MRI activity | Up to Week 48
Number of participates that are Anti JCV antibody positive at baseline | At Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (11):
- Russia (11):
  - Research Site, Belgorod
  - Research Site, Kaluga
  - Research Site, Kazan'
  - Research Site, Krasnodar
  - Research Site, Kursk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Perm
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Smolensk